CLINICAL TRIAL: NCT00199212
Title: A Phase I, Open Label, Dose-escalating Study of the Proteasome Inhibitor PS-341 in Combination With Two Schedules of Herceptin, in Patients With Advanced Breast Cancer That Overexpresses HER-2
Brief Title: PS-341 in Combination With Herceptin in Advanced Breast Cancer That Overexpresses HER-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Dr Fatima Cardoso, Institut Jules Bordet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Herceptin-proteasome inhibitor
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Carcinoma Breast Stage IV
Keywords: HER-2 positive; metastatic breast cancer patients
MeSH Terms: conditions — Breast Neoplasms | interventions — Bortezomib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Combination of trastuzumab and PS-341 — Trastuzumab and velcade are used according standard procedure
  Other Names: PS-341, velcade; trastuzumab, herceptine

SUMMARY:
The main objective of this study is to determine the feasibility of the combination of the proteasome inhibitor bortezomib (PS-341, Velcade) with trastuzumab (Herceptin) and to determine the best dose of bortezomib to combine with two trastuzumab schedules, weekly and 3-weekly.

DETAILED DESCRIPTION:
Phase 1 study to determine the feasibility of the combination of the proteasome inhibitor bortezomib (PS-341, Velcade) with trastuzumab (Herceptin) given either weekly or 3-weekly.

Additionally, hints about efficacy of the combination will be looked upon.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender
2. Age >= 18 years
3. ECOG performance status < 2
4. Histologically proven diagnosis of breast cancer
5. Locally advanced and/or metastatic disease
6. Life expectancy of three months or longer
7. No concurrent second malignancy (except for adequately treated basal cell carcinoma of the skin, in situ carcinoma of the cervix or contralateral breast cancer). Any prior second malignancy must be in remission for >= 5 years (except for contralateral breast cancer).
8. No other serious illness or medical condition including:

   * History of documented congestive heart failure; angina pectoris requiring antianginal medication; evidence of recent (< 6 months) transmural infarction on electrocardiogram (ECG); poorly controlled hypertension (e.g. systolic > 180 mmHg or diastolic greater than 100 mmHg); clinically significant valvular heart disease; or high-risk uncontrolled arrhythmias.
   * Chronic lung disease
   * History of significant neurological or psychiatric disorders that would prohibit the understanding and giving of informed consent, including psychotic disorders, mental retardation, and dementia.
   * Active concurrent infection
9. No symptomatic central nervous system (CNS) metastases
10. No rapidly progressive visceral metastases requiring immediate chemotherapy
11. No concurrent anti-cancer treatment is allowed.
12. Prior investigational biological agents are allowed, with the exception of anti-HER-2 therapy for any reason.
13. Previous hormonal therapy is allowed, as adjuvant and/or for metastatic breast cancer (MBC).
14. Adjuvant and MBC chemotherapy allowed, provided that a minimum of 4 weeks interval has elapsed between last chemotherapy administration and first study drug dose. All patients who, in the opinion of the investigator, could benefit from single agent Herceptin® and are not considered suitable for treatment with chemotherapy plus Herceptin® can be considered for this protocol.
15. A maximum cumulative dose of previous doxorubicin < 360 mg/m2 or a maximum cumulative dose of epirubicin < 720 mg/m2
16. Concomitant use of bisphosphonates is allowed, however if bisphosphonates are started during the trial for worsening bone pain, patients should be assessed for possible progressive disease.
17. Adequate organ function as defined by:

    * Neutrophils >= 1.5 x 10^9/L
    * Platelets >= 100 x 10^9/L
    * Bilirubin <= 1.5 x upper limit of normal (ULN)
    * Transaminases <= 2.5 x ULN or <= 5 x ULN if liver metastasis
    * Creatinine <= 1.5 x ULN
18. Overexpression of HER-2 in the invasive component of the primary tumor, according to one of the following definitions:

    * 3+ overexpression by immunohistochemistry (IHC) or
    * 2+ overexpression by IHC and fluorescence in situ hybridization (FISH) test demonstrating c-erbB2 gene amplification (ratio of c-erbB2 gene signals to centromere 17 signals > 2)
19. Baseline left ventricular ejection fraction (LVEF) > 50% measured by multiple gated acquisition scan (MUGA) or echocardiography
20. Evaluable or uni-dimensionally measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
21. Women of childbearing potential must have a negative serum or urine pregnancy test and be willing to use acceptable methods of birth control.
22. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
23. Before patient registration/randomization, informed consent must be given according to International Conference of Harmonization/European Union Good Clinical Practice (ICH/EU GCP), and national/local regulations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and maximum tolerated dose | before recurrence
  Combination of Velcade and Herceptine in breast metastatic patients
Time of recurrence | time of recurrence
  safety and tolerability of combinaison before recurrence of metastatic breast cance

SECONDARY OUTCOMES:
Response rate | time before response rate
  Tolerability and safety of combination of velcade and Herceptine

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Cardoso, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium